CLINICAL TRIAL: NCT03836183
Title: Interest of Pleuropulmonary Ultrasound Associate With Clinical Examination to Check the Good Position of the Double Lumen Tube Intubation in Patients Undergoing Thoracic Surgery
Brief Title: Pleuropulmonary Ultrasound With Clinical Examination to Check the Good Position of the Double Lumen Tube Intubation
Acronym: Echo-Thorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Pro-arte (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2018-EchoThorax
Record Dates: First submitted 2019-01-04; First posted 2019-02-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Thoracic; Surgery
Keywords: bronchoscopy; ultrasound; thorax
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound (Other): * ultrasound is the only study group for all the patients
  * pleuropulmonary ultrasound
  * clinical examination
  * fibroscopy.
  Interventions: Diagnostic Test: Pleuropulmonary ultrasound with clinical examination

INTERVENTIONS:
Diagnostic Test: Pleuropulmonary ultrasound with clinical examination — Pleuropulmonary ultrasound associate with a clinical examination

SUMMARY:
Using a new ultrasound approach, allow us to avoid the systematic use of bronchoscopy which is an invasive procedure. Although rare, several complications are known with, among other things, the occurrence of pulmonary infections, pneumothorax associated with increased pressure in the airways, atelectasis or bronchospasm.

Avoid the systematic control by fibroscopy in simple cases which makes it possible to overcome the complications related to its use and its cost.

The investigators want to evaluate the diagnostic value of the echographic strategy in 2 steps (2D and TM) on 3 sections (pulmonary field on the axillary line of the 2 sides and left upper lobe) associated with the clinical examination in preoperative by comparing with the gold standard: fibroscopy. Clinical examination and pleuropulmonary ultrasound should have a positive predictive value of at least 85%.

DETAILED DESCRIPTION:
In thoracic surgery, it is common to use selective intubation probes to exclude from ventilation the lung operated by the surgeon. It is recommended to perform a bronchoscopy which is the reference examination to confirm the good position of these probes. The interest of systematically controlling the good position of the left selective intubation probe by fibroscopy is controversial.

The interest of ultrasound for the diagnosis of pleuro-pulmonary pathologies is certain in resuscitation and emergency context for the diagnosis of pneumothorax, haemothorax and atelectasis.

The use of pleuropulmonary ultrasound in anesthesiology is the subject of studies. Several teams used it to ensure proper endotracheal tube positioning and to diagnose selective intubation. In fact, it has been shown that to control the position of the probe more precisely, ultrasound is more efficient than auscultation.

The aim of this work is to show by a large-scale prospective study that pleuropulmonary ultrasound associated with the clinical examination confirms the exclusion of the operated lung. the absence of systematic control of the positioning of the probe by fibroscopy allow financial gain and a reduction in the risk of morbidity related to the realization of this invasive gesture.

ELIGIBILITY:
Inclusion Criteria:

* Patient will benefit from thoracic or cardiac surgery requiring selective left intubation.
* Affiliation to the French social security

Exclusion Criteria:

* Minor patients
* Refusal of the patient
* Patients under guardianship, curators.
* Surgery not compatible with a visualization of the pleural slip in echography: surgery of pneumothorax or liquid effusion
* History likely to disturb the detection of pleural slip on ultrasound: pneumothorax surgery
* Predictable intubation difficulties and the need for selective bronchial blocker intubation
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of the clinical examination associated with pleuropulmonary ultrasound in order to diagnose the correct exclusion of the operated lung in thoracic surgery. | During peroperative period
  The presence of all these following data makes it possible to qualify the exclusion as correct. Clinical data collected : absence of vesicular murmur at the auscultation, absence of leaks (less than 10% or insufflation pressures < 4kPa (kilopascal) for a volume of 4 -5ml / kg in spirometry, and absence of bubbles in the bubble test. Ultrasound data collected: absence of pleural slip in 2D mode, presence of the bar code sign in TM mode.

SECONDARY OUTCOMES:
to evaluate the diagnostic performance of pleuropulmonary ultrasound alone to diagnose the right exclusion of the operated lung in thoracic surgery. | During peroperative period
  Only the presence of the two following non metric imaging criteria makes it possible to qualify the exclusion as correct. Ultrasound criteria : absence of pleural sliding in 2D mode, Presence of the bar code sign in TM mode.
To evaluate the interobserver validity of pleuropulmonary ultrasound as a diagnostic test for pulmonary exclusion. | at the end of the inclusion period, an average of 1 year
  Number of participant with the presence of the two following non metric imaging criteria makes it possible to qualify the lung exclusion as correct. Ultrasound criteria : absence of pleural sliding in 2D mode, Presence of the bar code sign in TM mode. Evaluation on ultrasonographic loops blinded registered from bronchoscopy diagnosis.
Assess the surgeon's satisfaction with lung exclusion: visual analogue scale | at the end of the surgery, day 1
  Quantified satisfaction scale in visual analogue scale. (from 0: worse outcome, to 10: better outcome)
determination of the performance of color Doppler in the diagnosis of pulmonary exclusion, visually assessed by presence of colour. | During ultrasound
  absence or presence of color in the pulmonary parenchyma on the 3 movements (pulmonary fields on the axillary line of the 2 sides and left upper lobe). The absence of color corresponding to a correct exclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Alabaladejo Pierre, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Chu grenoble alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No